CLINICAL TRIAL: NCT00186121
Title: A Phase II Trial of Arimidex Plus Zoladex in the Treatment of Hormone Receptor Positive, Metastatic Carcinoma of the Breast in Premenopausal Women
Brief Title: Estradiol Suppression for the Treatment of Metastatic Breast Cancer in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Melinda Telli, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13429; 75597 (Other: Stanford IRB alternate); BRSMTS0001 (Other: OnCore); 1033VS0012 (Other: alternate)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anastrozole + Goserelin (Experimental): Participants received goserelin 3.6 mg subcutaneously monthly. Beginning on Day 22 after the first dose of goserelin, participants began taking anastrozole 1 mg orally daily. No dose attenuation or escalation was allowed for either goserelin or anastrozole.
  Interventions: Drug: Anastrozole (Arimidex); Drug: Goserelin (Zoladex)

INTERVENTIONS:
Drug: Anastrozole (Arimidex) — Anastrozole is a prescription hormonal treatment that helps fight breast cancer by lowering the amount of estrogen in the body. It is a non-steroidal aromatase inhibitor, which significantly lowers serum estradiol (estrogen) concentrations, without interfering with the formation of adrenal corticosteroids or aldosterone
  Other Names: Arimidex
Drug: Goserelin (Zoladex) — Goserelin is a palliative treatment of advanced breast cancer in pre- and perimenopausal women
  Other Names: Zoladex

SUMMARY:
To evaluate the antitumor activity, toxicity, and effectiveness of the combination of goserelin (Zoladex) and anastrozole (Arimidex) in the treatment of premenopausal women with hormone receptor positive metastatic carcinoma of the breast.

DETAILED DESCRIPTION:
Pre-menopausal women with estrogen and/or progesterone receptor positive, metastatic or recurrent breast cancer were enrolled and treated with goserelin (Zoladex) monthly and began anastrozole (Arimidex) daily for 21 days following the first injection of goserelin. Participants continued on treatment until disease progression or unacceptable toxicity.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-confirmed, bi-dimensionally measurable, recurrent or metastatic carcinoma of the breast that is progressive
* Premenopausal, defined as any of:

  1. Last menstrual period within 3 months, or
  2. Post-hysterectomy without bilateral oophorectomy and with follicle-stimulating hormone (FSH) in the premenopausal range, or,
  3. If tamoxifen administered within the past 3 months, plasma estradiol must be in the premenopausal range
* Either positive estrogen and/or progesterone receptor determination by Immunohistochemistry (IHC) or competitive binding assay on metastatic disease, or if not performed on their metastatic disease a positive result on their primary breast cancer specimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Granulocytes > 1500/mm^3
* Platelets > 100,000/mm^3
* Serum glutamic oxaloacetic transaminase (SGOT) < 2.5 x upper limit of normal
* Total bilirubin < 1.5 mg/dL
* May have received irradiation to bony sites of disease for pain control or for prevention of fracture. The irradiated site(s) will NOT be evaluable for disease response.
* Must be using effective contraception or not be of childbearing potential
* Signed written informed consent

INCLUSION CRITERIA

* Active, unresolved infection
* Active malignancy other than breast cancer, in situ carcinoma of the cervix, or non-melanomatous skin cancers in the past 5 years
* Prior treatment with an aromatase inhibitor or inactivator
* Prior treatment with an luteinizing hormone-releasing hormone (LH/RH) agonist/antagonist
* Adjuvant chemotherapy within 6 months of study entry.
* Received chemotherapy or hormonal therapy in the 3 weeks prior to enrollment
* Central nervous system metastasis
* Lymphangitic pulmonary metastasis
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Telli, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carlson RW, Theriault R, Schurman CM, Rivera E, Chung CT, Phan SC, Arun B, Dice K, Chiv VY, Green M, Valero V. Phase II trial of anastrozole plus goserelin in the treatment of hormone receptor-positive, metastatic carcinoma of the breast in premenopausal women. J Clin Oncol. 2010 Sep 1;28(25):3917-21. doi: 10.1200/JCO.2009.24.9565. Epub 2010 Aug 2. PMID 20679610

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anastrozole + Goserelin
Started (Consented) | 35
Completed | 32
Not Completed | 3
Not completed — Subject withdrawal (no treatment) | 1
Not completed — Underwent oophorectomy (no treatment) | 1
Not completed — Not eligible (no treatment) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 43 [28 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was determined as the sum of the Complete Response (CR) rate + Partial Response (PR) rates.
  * CR = Complete disappearance of all clinically- or pathologically-detectable malignant disease for at least 4 weeks.
  * PR = ≥ 50% decrease in tumor size for at least 4 weeks, without any new lesion or any ≥ 25% increase in size of any lesion.
  All measurements by ruler or calipers.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anastrozole + Goserelin: Participants received goserelin 3.6 mg subcutaneously monthly. Beginning on Day 22 after the first dose of goserelin, participants began taking anastrozole 1 mg orally daily.
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
percentage of participants | 37.5 [21 to 56]

2. Secondary Outcome: Clinical Benefit Rate
Description: The overall clinical benefit rate of goserelin followed by anastrozole was evaluated, as determined as the sum of the Complete Response (CR) rate + Partial Response (PR) rate + Stable Disease (SD) rate.
  * CR = Complete disappearance of all clinically- or pathologically-detectable malignant disease for at least 4 weeks.
  * PR = ≥ 50% decrease in tumor size for at least 4 weeks, without any new lesion or any ≥ 25% increase in size of any lesion.
  * SD = No significant change in measurable or evaluable disease for at least 4 weeks.
  All measurements by ruler or calipers.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
percentage of participants | 71.9 [53 to 86]

3. Secondary Outcome: Response Rates
Description: The numbers of participants with metastatic breast cancer experiencing Complete Response (CR); Partial Response (PR); or Stable Disease (SD) after treatment with goserelin followed by anastrozole are reported.
  * CR = Complete disappearance of all clinically- or pathologically-detectable malignant disease for at least 4 weeks.
  * PR = ≥ 50% decrease in tumor size for at least 4 weeks, without any new lesion or any ≥ 25% increase in size of any lesion.
  * SD = No significant change in measurable or evaluable disease for at least 4 weeks.
  All measurements by ruler or calipers.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 11
  Stable Disease (SD) | 11

4. Secondary Outcome: Time-to-Progression (TTP)
Description: Time-to-progression (TTP) was assessed as the median observed in the participant group.
  Progression of disease was considered, per protocol, to be ≤ 25% increase in the area of any malignant lesion greater than 2 square cm, or ≤ 25% increase in the sum of the products of the longest perpendicular diameters of individual lesions in a given organ, when compared to baseline values or after therapeutic response.
Time Frame: up to 63 months
Measure: Median (Full Range); unit: months
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
months | 8.3 [2.1 to NA] — The upper limit of the range for TTP was not determined / not reached.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as the median observed in the participants receiving goserelin followed by anastrozole.
Time Frame: up to 63 months
Measure: Median (Full Range); unit: months
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
months | NA [11.1 to NA] — The median and upper limit of the range for OS were not reached / not determined. The upper limit exceeded 63 months.

6. Secondary Outcome: Estradiol Suppression
Description: Plasma estradiol determinations were performed at baseline, 1 month, 3 months, and 6 months using the Coat-A-Count Estradiol competitive binding assay system, which has a calibrated range for estradiol of 20 to 3,600 pg/mL with an analytical sensitivity of 10 pg/mL.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL estradiol
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
pg/mL estradiol
  Mean at Baseline | 74.7 (NA) — The study manuscript is the only source of these results data. The location of original study files is not known. The original data values are not available. Only the mean value without dispersion is known. No measure of dispersion is available.
  Mean at 1 month treatment | 20.8 (NA) — The study manuscript is the only source of these results data. The location of original study files is not known. The original data values are not available. Only the mean value without dispersion is known. No measure of dispersion is available.
  Mean at 3 months treatment | 18.7 (NA) — The study manuscript is the only source of these results data. The location of original study files is not known. The original data values are not available. Only the mean value without dispersion is known. No measure of dispersion is available.
  Mean at 6 months treatment | 14.8 (NA) — The study manuscript is the only source of these results data. The location of original study files is not known. The original data values are not available. Only the mean value without dispersion is known. No measure of dispersion is available.

7. Secondary Outcome: Serious Adverse Events
Description: The toxicity of the treatment regimen of goserelin followed by anastrozole is estimated by the rate of Serious Adverse Events (SAEs) that occurred during the course of the study.
Time Frame: 6 months
Measure: Number; unit: Serious Adverse Events (SAEs)
Arm/Group | Anastrozole + Goserelin
Number analyzed (Participants) | 32
Serious Adverse Events (SAEs) | 0

ADVERSE EVENTS:
Time Frame: Up to 63 months
Arm/Group | Anastrozole + Goserelin
All-Cause Mortality (participants affected / at risk) | 15/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 32/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole + Goserelin (N=32)
Hot flush (Vascular disorders) | 19 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (17)
Fatigue (General disorders) | 16 (16)
Headache (Nervous system disorders) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Neuropathy (Nervous system disorders) | 6 (6)
Vaginal dryness (Reproductive system and breast disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Mood alteration (Psychiatric disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
General disorders, other: Increased Sweating (General disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Gastrointestinal disorders - Other, cramping (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Heart burn (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No